CLINICAL TRIAL: NCT06610487
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of FT1 in Healthy Adult Volunteers
Brief Title: A Study of FT1 in Healthy Adult Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Peg-Bio Biopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQPJ-FT1-001
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Diarrhea Caused by Drug (Disorder)
Keywords: Chemotherapy induced diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Single-dose FT1 (Experimental): A single dose of FT1 will be administered, subcutaneous injection
  Interventions: Drug: FT1
- Single-dose FT1 Placebo (Placebo Comparator): A single dose of FT1 Placebo will be administered, subcutaneous injection
  Interventions: Drug: Placebo
- Multiple-dose FT1 (Experimental): FT1 will be administered once weekly for 3 weeks, subcutaneous injection
  Interventions: Drug: FT1
- Multiple-dose FT1 Placebo (Placebo Comparator): FT1 Placebo will be administered once weekly for 3 weeks, subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FT1 — Six dose levels will be evaluated in single-dose part, and three dose levels in multiple-dose part.
  Arms: Multiple-dose FT1; Single-dose FT1
Drug: Placebo — Placebo will be administered.
  Arms: Multiple-dose FT1 Placebo; Single-dose FT1 Placebo

SUMMARY:
The main aim of this clinical trial is to assess the safety of FT1 in participants aged 18 to 45 years. The main questions it aims to answer are:

• Is FT1 safe in healthy adults? Researchers will compare FT1 to a placebo (a look-alike substance that contains no drug) to see if FT1 is safe and active in human.

Participants will

* Receive one subcutaneous injection or multiple injections of FT1 or placebo according to weight.
* Visit the clinic for assessment.

DETAILED DESCRIPTION:
This study is a first-in-human study, which is a single-center, randomized, placebo-controlled, double-blind, dose escalation clinical study, aiming to evaluate the safety, tolerability, pharmacokinetics and immunogenicity of FT1 in healthy adult volunteers.

The trial is divided into 2 parts, single-dose part and multiple-dose part. In multiple-dose part, participants will receive once weekly subcutaneous injection of FT1 for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. healthy male or female subjects aged 18 to 45 years (inclusive);
2. Male subjects weighing ≥ 50.0kg, female subjects weighing ≥ 45kg; body mass index (BMI) in the range of 19.0-26.0 kg/m^2 (inclusive);
3. Voluntarily participate and sign the informed consent form;
4. Be able to complete the trial in accordance with the protocol.

Exclusion Criteria:

1. History of allergic diseases (including but not limited to asthma, urticaria, allergic rhinitis), or a history of drug allergies, or a history of allergies to the ingredients of the investigational drug;
2. Abnormal results of vital signs, physical examination, 12 lead electrocardiogram examination, and laboratory tests (including blood routine, urine routine, blood biochemistry, coagulation function, thyroid function) during the screening period with clinically significance determined by the researcher;
3. History or experiencing diseases with abnormal clinical manifestations, including but not limited to neurological/psychiatric, respiratory, cardiovascular, digestive, blood and lymphatic, urinary, endocrine, immune system diseases, or any other diseases or physiological conditions that may interfere with test results;
4. With intestinal polyp disease or have undergone intestinal polyp surgery within 6 months before screening;
5. Any positive results of hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody and treponema pallidum (TP) antibody test;
6. Positive urine test results for drug abuse (including morphine, methamphetamine, ketamine, cocaine, methylenedioxymethamphetamine, tetrahydrocannabinolic acid);
7. History of drug use or drug abuse (including the use of prohibited substances for medical use and controlled drugs);
8. History of critical surgery within 3 months before screening or plan to undergo surgery during the trial, as well as a history of surgery that may affect drug absorption, distribution, metabolism and excretion;
9. Participated in any clinical trial as a subject within 3 months before screening;
10. Have donated blood or lost more than 400 mL of blood/plasma within 3 months before screening (except for physiological blood loss in women);
11. Alcoholics (i.e. males drinking more than 28 standard units of alcohol per week and females drinking more than 21 standard units of alcohol per week, with 1 standard unit containing 14g of alcohol, such as 360mL beer or 45mL of 40% spirits or 150mL wine) or those who have frequently consumed alcohol within the previous 6 months (i.e. drinking more than 14 standard units of alcohol per week), or those who cannot abstain from alcohol during the trial, or those who have a positive alcohol breath test;
12. Took any prescription or over-the-counter drugs, as well as any functional vitamins or herbal products within 14 days before screening;
13. Have a long-term history of excessive consumption of tea, coffee or caffeinated beverages (more than 8 cups per day, 1 cup = 250mL)
14. Smoked more than 5 cigarettes per day within 6 months before screening;
15. Cannot guarantee to refrain from strenuous exercise, smoking and special diet (including grapefruit, chocolate, tea, cola, or any food or beverage containing caffeine, alcoholic beverages or other food or beverage that affects drug absorption, distribution, metabolism and excretion) from 48 hours before medication to the last blood collection;
16. Pregnant or lactating women, or female subjects who have had unprotected sex in the past two weeks, or female subjects with positive pregnancy test; subjects (or their partners) who have fertility plans or sperm/egg donations during the entire trial period and within 6 months after the last medication, and are unwilling to take one or more contraceptive measures during the trial and within 6 months after the last medication;
17. Cannot tolerate venous puncture or have difficulty in venous blood collection;
18. History of needle phobia or blood phobia or known severe bleeding tendency;
19. Have special dietary requirements and cannot follow a uniform diet;
20. The investigator believes the subject is unsuitable for participating in this clinical study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-03-06 (Estimated); Study Completion 2025-05-06 (Estimated)

PRIMARY OUTCOMES:
Treatment-related Adverse Events | up to 29 days in single-dose part, and up to 43 days in multiple-dose part
  To evaluate the adverse events as characterized by type, frequency, severity as graded by the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, timing, seriousness, and relationship to study therapy after administration.

SECONDARY OUTCOMES:
The Area Under the Curve from dosing to the time of the last measured concentration (AUC0-t) | up to 29 days in single-dose part, and up to 43 days in multiple-dose part
  Pharmacokinetic parameter
Maximum plasma concentration (Cmax) | up to 29 days in single-dose part, and up to 43 days in multiple-dose part
  Pharmacokinetic parameter
The half-life (t1/2) | up to 29 days in single-dose part, and up to 43 days in multiple-dose part
  Pharmacokinetic parameter
Anti-drug Antibody | up to 29 days in single-dose part, and up to 43 days in multiple-dose part
  Immunogenicity of FT1

CONTACTS AND LOCATIONS:
Locations (1):
- Bishan Hospital of Chongqing, Chongqing, Chongqing Municipality, China